CLINICAL TRIAL: NCT06123117
Title: Single Transversus Abdominis Laparoscopy-guided Plane Block Combined With Local Trocar Site Ropivacaine Infiltration (STALL) vs Sole Local Wound Infiltration in LCC (Laparoscopic CholeCystectomy) - Double-blinded Randomized Controlled Trial.
Brief Title: STALL vs Sole Local Wound Infiltration in Laparoscopic Cholecystectomy
Acronym: STALL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Roman Kornosev, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 7351
Record Dates: First submitted 2023-11-05; First posted 2023-11-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Cholelithiasis; Cholecystitis; Gallbladder Cancer
Keywords: laparoscopic transversus abdominis plane block
MeSH Terms: conditions — Cholelithiasis; Cholecystitis; Gallbladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients are analyzed following the intention to treat in three subgroups:
  1. Patients treated in "day-care" outpatient surgical unit (DS): TAP+local vs local.
  2. Patients treated electively in the inpatient surgery unit (IS): TAP+local vs local.
  3. Emergency surgery patients (ES): TAP+local vs local.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be blinded to patients and recovery room personnel, as well as the ward nurses and physicians, but not to operating surgeon(s), anesthesiologist(s), and nurses, treating patients during the surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Daycare: STALL (Experimental): Local ropivacaine infiltration + laparoscopically controlled TAP (transversus abdominis plane block). Daycare patients.
  Interventions: Procedure: single transversus abdominis laparoscopy-guided plane block; Procedure: local trocar site ropivacaine infiltration
- Daycare: local only (Active Comparator): Local ropivacaine infiltration only. Daycare patients.
  Interventions: Procedure: local trocar site ropivacaine infiltration
- In-patient: STALL (Experimental): Local ropivacaine infiltration + laparoscopically controlled TAP. In-patient surgery.
  Interventions: Procedure: single transversus abdominis laparoscopy-guided plane block; Procedure: local trocar site ropivacaine infiltration
- In-patient: local only (Active Comparator): Local ropivacaine infiltration only. In-patient surgery.
  Interventions: Procedure: local trocar site ropivacaine infiltration
- Emergency: STALL (Experimental): Local ropivacaine infiltration + laparoscopically controlled TAP. Emergency patients.
  Interventions: Procedure: single transversus abdominis laparoscopy-guided plane block; Procedure: local trocar site ropivacaine infiltration
- Emergency: local only (Active Comparator): Local ropivacaine infiltration only. Emergency patients.
  Interventions: Procedure: local trocar site ropivacaine infiltration

INTERVENTIONS:
Procedure: single transversus abdominis laparoscopy-guided plane block — please see arm/group descriptions
  Other Names: STALL
  Arms: Daycare: STALL; Emergency: STALL; In-patient: STALL
Procedure: local trocar site ropivacaine infiltration — please see arm/group descriptions

SUMMARY:
This trial is a prospective randomized superiority trial comparing sole ropivacaine based local trocar site infiltration to local infiltration combined with laparoscopic ropivacaine TAP block (STALL) in LCC.

There are only a few randomized trials comparing sole local anesthesia to additional laparoscopic TAP block in laparoscopic cholecystectomy and they have yet failed to show evidence in favor of TAP block.

We hypothesize STALL (Single Transversus Abdominis Laparoscopy-guided plane block combined with Local trocar site ropivacaine infiltration) is superior to local port site infiltration, provided that the sample size is sufficiently big.

The aim of this randomized study is to compare the efficacy of sole local anesthesia of trocar sites to STALL in LCC.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for elective or emergency LCC, aged over 18 and able to give an informed consent.

Exclusion Criteria:

* Age under 18 years, chronic daily opioid and/or pain tolerance / pain threshold -modifying medication use (abuse), pregnancy, known allergy to local anesthetics, diagnosed severe coagulopathy and incapability to give informed consent for whatever reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
cumulative opioid consumption during the stay at the recovery | duration of stay at the recovery (estimated 1-4 hours)
  all groups; mg, morphine equivalent

SECONDARY OUTCOMES:
maximum NRS score during the day of surgery, after discharge (daycare / outpatient) | 30 min after surgery, every 60 min afterwards; 2 days
  NRS (Numerical Rating Scale): 0-10
cumulative opioid consumption (emergency and inpatient surgery) | while admitted; est. 2 days
  mg, morphine equivalent

OTHER OUTCOMES:
maximum NRS score during the stay at the recovery | until the patient is either discharged to ward or home (day surgery patients), est. 1-4 hours
  0-10
average NRS score during the stay at the recovery | duration of stay at the recovery, est. 1-4 hours
  0-10
NRS score in multiple time points | every hour until discharge and at discharge = "ready to go" / "ready for transfer" (during in-hospital care), est. 48 hours
  if awake
procedure time | minutes; est. 60 - 180 minutes
  min
time necessary in recovery room | minutes; est. 60 - 260 min
  min, (= "patient ready to be discharged" timestamp OR "patient ready for transfer")
complications related to the use of local anesthetics | est. 0 - 7 days
  TAP + port site infiltration complications (as per trial plan) + other complications according to Clavien-Dindo classification
patient general satisfaction with pain management | prespecified: about 4 hours, 2 days, 7 days, 30 days
  using questionnaires, multiple timepoints: recovery stay, hospital stay, discharge, feedback after 7 days
time from surgery to discharge | est. 2 - 48 hours
  min
number of patients contacting the hospital regarding inadequate pain management | after discharge and before day 30
  n
prevalence of postoperative nausea and vomiting (PONV) and difference in subgroups | est. 0 - 4 (8) hours
  n; %
difference in NRS (if any) between patients received remifentanil or fentanyl intraoperatively | 0 - 4 hours
  delta
difference in NRS (if any) between patients received propofol or sevoflurane maintenance. | 0- 4 hours
  delta
pain-control failure & possible causes | acute: 0 - 2 days; chronic: t+30 days
  APS (acute pain service) contact, admission of DS subgroup patient to the ward due to pain, failure to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Henna Sammalkorpi, MD, PhD, Study Director — Helsinki UCH; Hanna Lampela, MD, PhD, Study Director — Helsinki UCH; Jukka Harju, MD, PhD, Doc, Study Director — Helsinki UCH
Locations (1):
- Jorvi hospital / HUS, Espoo, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siriwardana RC, Kumarage SK, Gunathilake BM, Thilakarathne SB, Wijesinghe JS. Local infiltration versus laparoscopic-guided transverse abdominis plane block in laparoscopic cholecystectomy: double-blinded randomized control trial. Surg Endosc. 2019 Jan;33(1):179-183. doi: 10.1007/s00464-018-6291-0. Epub 2018 Jun 25. PMID 29943054
- [Background] Bumblyte V, Rasilainen SK, Ehrlich A, Scheinin T, Kontinen VK, Sevon A, Vaaraniemi H, Schramko AA. Purely ropivacaine-based TEA vs single TAP block in pain management after elective laparoscopic colon surgery within an upgraded institutional ERAS program. Surg Endosc. 2022 May;36(5):3323-3331. doi: 10.1007/s00464-021-08647-z. Epub 2021 Sep 3. PMID 34480217
- [Background] Ruiz-Tovar J, Garcia A, Ferrigni C, Gonzalez J, Levano-Linares C, Jimenez-Fuertes M, Llavero C, Duran M. Laparoscopic-Guided Transversus Abdominis Plane (TAP) Block as Part of Multimodal Analgesia in Laparoscopic Roux-en-Y Gastric Bypass Within an Enhanced Recovery After Surgery (ERAS) Program: a Prospective Randomized Clinical Trial. Obes Surg. 2018 Nov;28(11):3374-3379. doi: 10.1007/s11695-018-3376-8. PMID 29980989
- [Background] Peng K, Ji FH, Liu HY, Wu SR. Ultrasound-Guided Transversus Abdominis Plane Block for Analgesia in Laparoscopic Cholecystectomy: A Systematic Review and Meta-Analysis. Med Princ Pract. 2016;25(3):237-46. doi: 10.1159/000444688. Epub 2016 Feb 16. PMID 26885872
- [Background] Breazu CM, Ciobanu L, Hadade A, Bartos A, Mitre C, Mircea PA, Ionescu D. The efficacy of oblique subcostal transversus abdominis plane block in laparoscopic cholecystectomy - a prospective, placebo controlled study. Rom J Anaesth Intensive Care. 2016 Apr;23(1):12-18. doi: 10.21454/rjaic.7518.231.obq. PMID 28913472
- [Background] Loizides S, Gurusamy KS, Nagendran M, Rossi M, Guerrini GP, Davidson BR. Wound infiltration with local anaesthetic agents for laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2014 Mar 12;2014(3):CD007049. doi: 10.1002/14651858.CD007049.pub2. PMID 24619479
- [Background] Elamin G, Waters PS, Hamid H, O'Keeffe HM, Waldron RM, Duggan M, Khan W, Barry MK, Khan IZ. Efficacy of a Laparoscopically Delivered Transversus Abdominis Plane Block Technique during Elective Laparoscopic Cholecystectomy: A Prospective, Double-Blind Randomized Trial. J Am Coll Surg. 2015 Aug;221(2):335-44. doi: 10.1016/j.jamcollsurg.2015.03.030. Epub 2015 Mar 27. PMID 25899736
- [Background] Tolchard S, Davies R, Martindale S. Efficacy of the subcostal transversus abdominis plane block in laparoscopic cholecystectomy: Comparison with conventional port-site infiltration. J Anaesthesiol Clin Pharmacol. 2012 Jul;28(3):339-43. doi: 10.4103/0970-9185.98331. PMID 22869941
- [Background] Ortiz J, Suliburk JW, Wu K, Bailard NS, Mason C, Minard CG, Palvadi RR. Bilateral transversus abdominis plane block does not decrease postoperative pain after laparoscopic cholecystectomy when compared with local anesthetic infiltration of trocar insertion sites. Reg Anesth Pain Med. 2012 Mar-Apr;37(2):188-92. doi: 10.1097/AAP.0b013e318244851b. PMID 22330261
- [Background] Bava EP, Ramachandran R, Rewari V, Chandralekha, Bansal VK, Trikha A. Analgesic efficacy of ultrasound guided transversus abdominis plane block versus local anesthetic infiltration in adult patients undergoing single incision laparoscopic cholecystectomy: A randomized controlled trial. Anesth Essays Res. 2016 Sep-Dec;10(3):561-567. doi: 10.4103/0259-1162.186620. PMID 27746552
- [Background] Ravichandran NT, Sistla SC, Kundra P, Ali SM, Dhanapal B, Galidevara I. Laparoscopic-assisted Tranversus Abdominis Plane (TAP) Block Versus Ultrasonography-guided Transversus Abdominis Plane Block in Postlaparoscopic Cholecystectomy Pain Relief: Randomized Controlled Trial. Surg Laparosc Endosc Percutan Tech. 2017 Aug;27(4):228-232. doi: 10.1097/SLE.0000000000000405. PMID 28472015
- [Background] Peng W, Huang S, Zhou S, Yang N, Zuo M. Case report: life-threatening coronary artery spasm under transversus abdominis plane block in combination with general anesthesia. BMC Anesthesiol. 2018 Oct 20;18(1):148. doi: 10.1186/s12871-018-0616-3. PMID 30342470
- [Background] Salaria ON, Kannan M, Kerner B, Goldman H. A Rare Complication of a TAP Block Performed after Caesarean Delivery. Case Rep Anesthesiol. 2017;2017:1072576. doi: 10.1155/2017/1072576. Epub 2017 Oct 29. PMID 29214081